CLINICAL TRIAL: NCT04190875
Title: Post-Discharge Growth and Development of Infants Who Received Targeted Fortification (High Versus Standard Protein Diet) in the NICU
Brief Title: Post-Discharge Growth and Development of Infants Who Received Targeted Fortification in the NICU
Status: Suspended | Type: Observational
Why Stopped: Inability to bring patients in for follow-up visits due to institutional restrictions related to COVID-19
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Amy Hair, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-44733
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Premature Infants
Keywords: Standard Protein Diet; High Protein Diet; Targeted Fortification; Post-Discharge Growth; Post-Discharge Body Compostion; Post-Discharge Neurodevelopment; Protein; Human Milk Diet; Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extremely low birth weight (ELBW) infants are at risk for slow growth, metabolic abnormalities, and poor neurodevelopmental outcomes. Postnatal growth standards are based on estimated intrauterine growth from historical cohort studies and post-mortem analyses. Despite current strategies aimed at appropriate nutrition, a large proportion of these infants have postnatal growth failure (anthropometric values < 10th percentile) reported in the literature as high as 89-99%. More recent data shows lower rates of postnatal growth failure but further improvement is still needed. Adequate growth is key to ensuring improved neurodevelopment and other outcomes.

The investigators are currently evaluating the effects of a high versus standard protein enteral diet on growth and body composition in infants less than or equal to 1000 grams birth weight in the Neonatal Intensive Care Unit. (H-38611). Infants less than or equal to 1000 grams birth weight are provided an enteral diet with a level of protein based on individual caloric and protein analysis of human milk also known as targeted fortification. The standard protein diet provides 3.5-3.8 g/kg/day of protein, while the high protein diet provides 4.2-4.5 g/kg/day.

The investigators have shown that infants who receive this diet achieve growth at targeted standards. As this diet is well tolerated and associated with improved outcomes in our highest risk neonates, it is imperative to evaluate the benefits of a high protein exclusive human milk diet and the possible positive changes in body composition, specifically lean mass, in these infants. Body composition in these infants receiving targeted fortification is being evaluated at 35-36 weeks post menstrual age.

Because these infants are at such high risk for poor growth and neurodevelopment, it is important to investigate the impact of a higher protein exclusive human milk diet on long-term neurodevelopmental outcomes, body composition, and growth at 18-24 months.

DETAILED DESCRIPTION:
The investigators plan to evaluate the effects of a high versus standard protein enteral diet utilizing targeted fortification on neurodevelopmental outcomes, growth, and body composition at 18-24 months in infants with a birth weight of less than or equal to 1000 grams.

Children who have completed a previous study (H-38611) evaluating the effects of a high versus standard protein diet utilizing targeted fortification with human donor milk products on weight, length, and body composition will be recruited for this study.

Infants in the previous study, (H-38611) were either born at Texas Children's Hospital or transferred to Texas Children's Hospital in the first 24 hours of life and admitted to our Neonatal Intensive Care Unit. These infants had a birth weight of less than or equal to 1000 grams and were randomized to receive a standard protein diet (3.5-3.8 grams of protein per kilogram of body weight- the amount of protein recommended for premature babies by the American Academy of Pediatrics ) or a high protein diet (4.2-4.5 grams of protein per kilogram of body weight- the amount of protein recommended for premature babies by the European Society of Paediatric Gastroenterolgy, Hepatology, and Nutrition). Infants in both groups received recommended clinical guidelines for protein.

While the previous study (H-38611) evaluated the effects of a high versus standard protein diet on weight, length and body composition prior to discharge from the Neonatal Intensive Care Unit, this study (H-44733) will assess if the amount of protein in the diet the infant received impacted growth, body composition, and neurodevelopment at 18-24 months of life.

For the study (H-44733), parents of patients who completed H-38611 will be consented prior to discharge from the Neonatal Intensive Care Unit. For patients who completed the previous study (H-38611) and have been discharged, the investigators will contact the parents by telephone. The investigators will mail a consent form to parents interested in having their child complete the follow-up study (H-44733) so they can review the consent form. Then, if they want to participate in the study, they will contact study staff to schedule an appointment. At the beginning of the appointment study staff will obtain informed verbal and written consent in order to conduct study visit.

This study includes an outpatient visit at 18-24 months corrected gestational age. At the visit, the investigators will obtain baseline anthropometric data, interim medical history, demographic and socioeconomic information, and nutrition history of the child since discharge (formula, human milk, vitamins, and medications). A registered dietitian will ask parents questions about the child's current diet.

Next, body composition will be measured by whole body dual energy x-ray absorptiometry or DXA scan. DXA scan is the current gold standard to provide lean and fat body mass and bone mineral content results. DXA is a way to measure bone mineral density, or the amount of calcium and other minerals in the bones.

In addition, a Neurodevelopmental Evaluation as part of standard follow-up for extremely low birth weight infants (The Bayley Scales of Infant and Toddler Development, 3rd Edition) will be completed. The Bayley Scales of Infant and Toddler Development is used mainly to assess the mental and motor development of infants and toddlers, ages 1-42 months. It will be administered by a pediatric developmental physician.

Results of evaluations will be given to parents and recommendations for follow-up will be made by the physician completing the evaluation.

No interventions are part of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Children born prematurely, with birth weight of less than or equal to 1000 grams
* Born at Texas Children's Hospital or transferred to the Neonatal Intensive Care Unit from another hospital in the first 24 hours of life
* Completed a previous study (H-38611) in which the child received targeted protein fortification with donor human milk products

Exclusion Criteria:

* Infants not previously enrolled in a previous study (H-38611) in the Neonatal Intensive Care Unit at Texas Children's Hospital
* Infants enrolled in but did not complete a previous study (H-38611) in the Neonatal Intensive Care Unit at Texas Children's Hospital

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 18-24 months corrected age, who participated in an earlier study H-38611. These children were either born at Texas Children's Hospital in the first 24 hours of life and admitted to our Neonatal Intensive Care Unit. These infants had a birth weight of less than or equal to 1000 grams and were randomized to receive a standard protein diet (3.5-3.8 grams of protein per kilogram of body weight) or a high protein diet (4.2-4.5 grams of protein per kilogram of body weight). Infants in both groups received recommended clinical guidelines for protein.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Linear growth measured using a pediatric stadiometer | 18-24 months corrected age
  Linear growth will be measured in centimeters (cm) at the time of the outpatient visit for DXA scan.

SECONDARY OUTCOMES:
Body composition measured by dual-energy x-ray absorptiometry (DXA) | 18-24 months corrected age
  The subject will be scanned once in infant mode and once in adult mode during the time of the outpatient visit.
Neurodevelopment will be measured by administration of The Bayley Scales of Infant and Toddler Development, 3rd Edition | 18-24 months corrected age
  A developmental pediatrician will administer The Bayley Scales of Infant and Toddler Development at the time of the outpatient visit. This assessment consists of a series of developmental play tasks and takes between 45-60 minutes to administer and derives a developmental quotient. The measure consists of five scales. Raw scores of successfully completed items are converted to scale scores and to composite scores. Low/high scores for each scale are as following: Cognitive (55-145), Language (47-153), Motor (46-154), Social-Emotional (55-145). Children who score low on this assessment are at risk for future developmental problems.

CONTACTS AND LOCATIONS:
Overall Officials: Amy B Hair, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (1):
- Baylor College of Medicine / Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hair AB, Peluso AM, Hawthorne KM, Perez J, Smith DP, Khan JY, O'Donnell A, Powers RJ, Lee ML, Abrams SA. Beyond Necrotizing Enterocolitis Prevention: Improving Outcomes with an Exclusive Human Milk-Based Diet. Breastfeed Med. 2016 Mar;11(2):70-4. doi: 10.1089/bfm.2015.0134. Epub 2016 Jan 20. PMID 26789484
- [Background] Hair AB, Blanco CL, Moreira AG, Hawthorne KM, Lee ML, Rechtman DJ, Abrams SA. Randomized trial of human milk cream as a supplement to standard fortification of an exclusive human milk-based diet in infants 750-1250 g birth weight. J Pediatr. 2014 Nov;165(5):915-20. doi: 10.1016/j.jpeds.2014.07.005. Epub 2014 Aug 15. PMID 25130571
- [Background] Hair AB, Hawthorne KM, Chetta KE, Abrams SA. Human milk feeding supports adequate growth in infants </= 1250 grams birth weight. BMC Res Notes. 2013 Nov 13;6:459. doi: 10.1186/1756-0500-6-459. PMID 24220185